CLINICAL TRIAL: NCT04841512
Title: A Placebo-controlled, Double-blind Evaluation of Safety, Tolerability, and Efficacy of XT-150 for the Treatment of Facet Joint Osteoarthritis Pain
Brief Title: Preliminary Safety and Efficacy of XT-150 in Facet Joint Osteoarthritis
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: COVID - Lack of recruitment
Sponsor: Xalud Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XT-150-1-0301
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Osteoarthritis, Spine
Keywords: gene therapy; non-viral plasmid; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Spine; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Unblinded pharmacy, blinded clinical staff for administration and assessments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator): Sterile phosphate-buffered saline for injection Single 1mL injection into the facet joint
  Interventions: Biological: XT-150
- XT-150 Dose #1 (Experimental): Lower dose of XT-150 sterile solution for injection Single 1 mL injection into the facet joint
  Interventions: Biological: XT-150
- XT-150 Dose #2 (Experimental): Higher dose of XT-150 sterile solution for injection Single 1 mL injection into the facet joint
  Interventions: Biological: XT-150

INTERVENTIONS:
Biological: XT-150 — non-viral Plasmid DNA encoding an IL-10 variant transgene

SUMMARY:
Preliminary safety and efficacy of XT-150 in the synovial capsule of osteoarthritic facet joints in the vertebra of the spine.

DETAILED DESCRIPTION:
This is a Phase 1, safety and efficacy study of XT-150 in adult participants experiencing back pain due to inflammation of the facet joint osteoarthritis (FJOA) and who are eligible for intra-synovial glucocorticoid injection, or radiofrequency ablation of medial branches of the primary dorsal ramus of the exiting nerve root, which innervates the adjacent facet joints.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, between 18 and 90 years of age, inclusive.
2. Sufficiently severe facet arthropathy (OA) of lumbar facets as determined by imaging, eg. CT or MRI, to establish an underlying basis of disease, as determined by usual bony and ligamentous signs of OA.
3. Complaint of nociceptive, mechanical pain of lumbar spine, in particular pain localized to paramedian axis as opposed to midline or radicular. Radicular pain as a secondary finding may be allowed if it is addition to mechanical pain and can be clinically distinguished by subject
4. Low Back Pain (LBP) worsened by activity or motion of region
5. Have had a positive diagnostic facet pain block with lignocaine; admittance if subject gains 50% relief of pain within 30 minutes of test injection
6. Be free of local or intra-articular infection, tumor or other causes of localized LBP, for example Including spondylolysis/pars defect, and adjacent vertebral body compression fracture based on MRI evaluation.
7. Symptomatic disease because of osteoarthritis, established by imaging of facet joint and defined as a worst pain of at least 40 at any time during the preceding week (based on scale of 0 to 100, with 100 representing "pain as bad as you can imagine") using Visual Analog Scale (VAS).
8. Stable analgesic regimen during the 4 weeks prior to enrollment.
9. Inadequate pain relief (minimum ≥50 mean on VAS with prior therapies lasting ≥3 months.
10. In the judgment of the Investigator, acceptable general medical condition
11. Male and female participants who are heterosexually active and not surgically sterile or post-menopausal must agree to use effective contraception, including abstinence, for the duration of the study and for 3 months after the study is completed
12. Have suitable facet joint anatomy for intra-articular injection
13. Willing and able to return for the follow-up (FU) visits
14. Able to reliably provide pain assessment (FAST test score R2≥0.7)
15. Able to read and understand study instructions, and willing and able to comply with all study procedures

Exclusion Criteria:

1. Hypersensitivity, allergy, or significant reaction to any ingredient of the study drug, including double-stranded DNA, mannose, and sucrose
2. Scheduled surgical procedure or nerve ablation to joint within the next 6 months; participant agrees not to schedule a surgical procedure, nerve ablation, or added facet injection within 6 months of study treatment
3. High peri-operative risks which in the judgment of the investigator preclude a safe facet joint injection procedure (e.g. extreme obesity putting injection accuracy at risk, etc.)
4. Current treatment with immunosuppressive (systemic corticosteroid therapy [equivalent to >10mg/day prednisone] or other strong immunosuppressant)
5. History of immunosuppressive therapy; high-potency systemic steroids in the last 3 months.
6. Currently receiving systemic chemotherapy or radiation therapy for malignancy
7. Clinically significant hepatic disease as indicated by clinical laboratory results ≥3 times the upper limit of normal for any liver function test (e.g., aspartate aminotransferase, alanine aminotransferase, lactate dehydrogenase)
8. Severe anemia (Grade 3; hemoglobin <8.0 g/dL, <4.9 mmol/L, <80 g/L; transfusion indicated), Grade 1 white cell counts (lymphocytes <LLN - 800/mm3; <LLN - 0.8 x 109 /L, neutrophils <LLN - 1500/mm3; <LLN - 1.5 x 109 /L)
9. Positive serology with reflex for human immunodeficiency virus, hepatitis B virus, or hepatitis C virus within 4 weeks of commencing the study
10. Significant neuropsychiatric conditions; dementia, major depression, or altered mental state that in the opinion of the Investigator will interfere with study participation
11. Current treatment with systemic antibiotics or antivirals (EXCEPTION: topical treatments)
12. Current treatment with anticoagulants, other than low-dose aspirin
13. Known or suspected history of active alcohol or intravenous/oral drug abuse within 1 year before the screening visit
14. Use of any investigational drug or device within 1 month before enrollment or current participation in a trial that included intervention with a drug or device; or currently participating in an investigational drug or device study.
15. Any condition that, in the opinion of the Principal Investigator, could compromise the safety of the participant, the participant's ability to communicate with the study staff, or the quality of the data

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | 6 months
  0 - 100, 100 worst possible pain

SECONDARY OUTCOMES:
Oswestry Disability Index | 6 months
  10 dimensions, 0 - 5 score in each, with 5 as worst score in a dimension

CONTACTS AND LOCATIONS:
Locations (1):
- Alfred Health, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
Not applicable. All patient records are de-identified